CLINICAL TRIAL: NCT03193203
Title: A Randomised, Open-label, Two-period, Two-sequence, Single-dose, Cross-over Study to Compare the Pharmacokinetics, Safety, and Tolerability of the Autoinjector and Pre-filled Syringe of SB4 in Healthy Male Subjects
Brief Title: Pharmacokinetics, Safety, and Tolerability Study of the Autoinjector and Pre-filled Syringe of SB4 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SB4-G12-NHV; 2016-004993-16 (EudraCT Number)
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): SB4 (etanercept) 50 mg/mL PFS and AI
  Interventions: Drug: Etanercept
- Sequence 2 (Experimental): SB4 (etanercept) 50 mg/mL AI and PFS
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — 50 mg/mL PFS and AI

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety, and tolerability of the autoinjector and pre-filled syringe of SB4 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18-55 years
* Have a body weight between 60.0 - 85.5 kg (inclusive) and a body mass index between 20.0 - 28.0 kg/m2 (inclusive)

Exclusion Criteria:

* Have a history and/or current presence of clinical significant atopic allergy, hypersensitivity or allergic reactions, also including known or suspected clinically relevant drug hypersensitivity to etanercept or to any of the excipient
* Have either active or latent TB or who have a history of TB
* Have clinically significant active infection within 4 weeks before the first IP administration
* Have had a history of serious infection
* Have previously been exposed to etanercept, if known
* Have previously been exposed to a biological agent or immunosuppressive agent within 120 days prior to the first IP administration
* Have a history of invasive systemic fungal infections or other opportunistic infections judged as relevant by the Investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-08-07 (Actual); Study Completion 2017-08-07 (Actual)

PRIMARY OUTCOMES:
AUCinf ACUinf | 56 days
  Area under the concentration-time curve from time zero to infinity
AUClast | 56 days
  Area under the concentration-time curve from time zero to the last quantifiable concentration
Cmax | 56 days
  Maximum serum concentration

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences, Groningen, Netherlands